CLINICAL TRIAL: NCT02954900
Title: Study of Web-based Decision Aids for Breast Cancer Risk Assessment and Increasing Breast Cancer Chemoprevention in the Primary Care Setting: Pilot
Brief Title: Know Your Risk: Assessment at Screening for Breast Cancer - Pilot Study
Acronym: KYRAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katherine D. Crew, Associate Professor of Medicine and Epidemiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAP4151 I; R01CA177995 (NIH)
Record Dates: First submitted 2016-07-12; First posted 2016-11-04 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer Prevention; Risk Assessment; Chemoprevention; Decision Making
MeSH Terms: conditions — Breast Neoplasms | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decision aid (Other): 50 women at high-risk for developing breast cancer will use a decision support tool, RealRisks, when discussing breast cancer risk with their providers who will have access to the BNAV provider clinical decision support tool.
  Interventions: Other: RealRisks; Other: BNAV

INTERVENTIONS:
Other: RealRisks — RealRisks is a web-based patient decision aid with modules that present information about risk assessment and chemoprevention.
  Other Names: RealRisks patient-centered decision aid (DA)
Other: BNAV — Breast Cancer Risk Navigation (BNAV) tool is a web-based decision support tool with modules that present pertinent information for primary care providers regarding breast cancer risk assessment and preventative measures for their patients.
  Other Names: Breast Cancer Risk Navigation (BNAV) tool; BNAV provider clinical decision support tool

SUMMARY:
The purpose of this pilot study is to evaluate a decision support website (RealRisks) designed to inform patients about breast cancer chemoprevention. It is coupled with a physician-centered (BNAV) decision support website as part of clinical workflow in the primary care setting. The investigator hypothesizes that improving accuracy of breast cancer risk perception and understanding of the risks/benefits of chemoprevention will enhance informed decision-making and uptake of breast cancer prevention strategies in the primary care setting.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among women in the U.S. and the primary prevention of this disease is a major public health issue. The U.S. Preventive Services Task Force and other professional organizations recommend that clinicians discuss chemoprevention with high-risk women. Breast cancer chemoprevention with anti-estrogens, such as tamoxifen, raloxifene, exemestane, and anastrozole, is under-utilized, despite several randomized controlled trials demonstrating a 40-65% decrease in breast cancer incidence among high-risk women. Compounding this underutilization is the fact that a large proportion of women may be unaware of their high-risk status due to the investigators inability to adequately screen them in the primary care setting. Further research is needed to determine how knowledge about breast cancer, actual/perceived risk, and risks/benefits of chemoprevention are best communicated to women in order to promote breast cancer prevention strategies.

This study assesses risk communication and shared decision-making in patient-clinician dyads by administering validated measures at baseline, after interacting with the tools prior to the clinic visit, and after the clinical visit (quantitative analysis); and by using observer-based methods of audio-tape recordings of their clinical encounters (qualitative analysis).

The investigator hypothesizes that combining a patient-centered decision aid with a physician-centered decision support tool integrated into clinic workflow will improve accuracy of breast cancer risk perception, facilitate referrals for specialized risk counseling, and increase chemoprevention uptake.

ELIGIBILITY:
Inclusion Criteria:

* 5-year breast risk of 1.67% or lifetime risk of 20% according to the Gail model
* The participant understands and is willing to provide informed consent in English or Spanish
* Has a primary care provider at Columbia University Medical Center (CUMC) / New York-Presbyterian Hospital

Exclusion Criteria:

* Prior use of a selective estrogen receptor modulator (SERM) or aromatase inhibitor (AI) for chemoprevention
* Prior history of breast cancer

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-15; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in the accuracy of risk perception (Likert Scale Score) | Baseline, 2 weeks
  To measure the patient's accuracy of perceived breast cancer risk before and after exposure to the RealRisks decision aid. Perception will be assessed by comparing the difference between a patient's perceived risk and their actual risk based on the Gail breast cancer model. Patients are asked to make a comparative risk assessment about themselves on a 3-point Likert scale.

SECONDARY OUTCOMES:
Change in a patient's breast cancer knowledge (Survey Score) | Baseline, 2 weeks
  To assess patient's breast cancer knowledge before and after exposure to the RealRisks decision aid by comparing the difference between a patient's responses to a 13-item scale assessing knowledge with response options of true, false, or unsure.
Chemoprevention uptake rate among high-risk women | 6 months
  To determine the uptake rate in the breast clinic after offering specialized risk counseling to a broader population of racially/ethnically diverse women screened in the primary care setting. Electronic health records will be used to track chemoprevention uptake after exposure to the RealRisks decision aid.
Referral rates to the breast clinic | 12 months
  To study appropriate referral rate by primary care providers of high-risk patients to the breast clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Crew, M.D., M.S., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kukafka R, Yi H, Xiao T, Thomas P, Aguirre A, Smalletz C, David R, Crew K. Why Breast Cancer Risk by the Numbers Is Not Enough: Evaluation of a Decision Aid in Multi-Ethnic, Low-Numerate Women. J Med Internet Res. 2015 Jul 14;17(7):e165. doi: 10.2196/jmir.4028. PMID 26175193
- [Background] Yi H, Xiao T, Thomas PS, Aguirre AN, Smalletz C, Dimond J, Finkelstein J, Infante K, Trivedi M, David R, Vargas J, Crew KD, Kukafka R. Barriers and Facilitators to Patient-Provider Communication When Discussing Breast Cancer Risk to Aid in the Development of Decision Support Tools. AMIA Annu Symp Proc. 2015 Nov 5;2015:1352-60. eCollection 2015. PMID 26958276
- [Derived] Kukafka R, Fang J, Vanegas A, Silverman T, Crew KD. Pilot study of decision support tools on breast cancer chemoprevention for high-risk women and healthcare providers in the primary care setting. BMC Med Inform Decis Mak. 2018 Dec 17;18(1):134. doi: 10.1186/s12911-018-0716-5. PMID 30558581